CLINICAL TRIAL: NCT04400734
Title: Esophagogastroduodenoscopy (EGD) is an Aerosol-generating Procedure: Proof of Concept Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2020.200
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Aerosol-generating Procedure, Esophagogastroduodenoscopy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, observational study — no intervention

SUMMARY:
The disease COVID-19 has been classified as pandemic by World Health Organisation (WHO) in March 2020. This poses a risk to healthcare workers. Whether esophagogastroduodenoscopy (EGD) is a aerosol-generating procedure (AGP) has brought controversy. Multiple international guidelines consider EGD as AGP based on expert consensus. No scientific data has been published regarding this. With a commercially available particle counter, we can differentiate the particle counts of different sizes in different areas of the endoscopy room. An increase from baseline particles of < 5um during or after the procedure would suggest that the procedure is an AGP. The baseline particle counts before and during the procedure are also recorded. The details of the procedure including procedure time and the use of sedation are also documented.

DETAILED DESCRIPTION:
The disease COVID-19 has been classified as pandemic by World Health Organisation (WHO) in March 2020. This poses a risk to healthcare workers. Whether esophagogastroduodenoscopy (EGD) is a aerosol-generating procedure (AGP) has brought controversy. Multiple international guidelines consider EGD as AGP based on expert consensus. No scientific data has been published regarding this. Currently, the term droplet is often taken to refer to droplets >5 microns (μm) in diameter that fall rapidly to the ground under gravity, and therefore are transmitted only over a limited distance (e.g. ≤1 m). In contrast, the term droplet nuclei refers to droplets ≤5 μm in diameter that can remain suspended in air for significant periods of time, allowing them to be transmitted over distances >1 metre. With a commercially available particle counter, we can differentiate the particle counts of different sizes in different areas of the endoscopy room. An increase from baseline particles of < 5um during or after the procedure would suggest that the procedure is an AGP. With the use of a commercial available particle counter, the number of particles of size (0.3um, 0.5um, 0.7um, 1um, 5um and 1um) are recorded. The baseline particle counts before and during the procedure are also recorded. The details of the procedure including procedure time and the use of sedation are also documented.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing EGD in the endoscopy unit of Prince of wales Hospital, Shatin, Hong Kong

Exclusion Criteria:

* EGD cannot be completed due to patient's condition
* Patients who are unstable and require extra medical attention
* Patients who refuse
* Patients who are not fit for consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing EGD in the endoscopy unit of Prince of wales Hospital, Shatin, Hong Kong will be included
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
The increase in particle counts of particle size (0.3um, 0.5um, 0.7um, 1um, 5um, 10um) during the procedure | during the procedure

SECONDARY OUTCOMES:
Procedure time | during the procedure
Use of sedation | during the procedure
Use of continuous suction | during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No